CLINICAL TRIAL: NCT02601716
Title: Clinical Trial of PfSPZ Vaccine Administered by Direct Venous Inoculation: Dose Optimization With Heterologous Challenge in Healthy Malaria-Naïve Adults
Brief Title: PfSPZ Vaccine: Dose Optimization With Heterologous Challenge in Healthy Malaria-Naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); University of Maryland (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Joint Warfighter Medical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMRC.2015.0009; CVD Malaria 26000 (Other: University of Maryland)
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine; Sporozoites; Controlled Human Malaria Infection
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — 1-acetyl-1,2,3,3a,8,8a-hexahydro-8a-hydroxy-5-methoxypyrrolo(2,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Experimental): Group 1 subjects (n=15) will receive 4 doses of PfSPZ Vaccine (4.5 x 10^5 PfSPZ/dose) every 2 days, followed by a single, boosting dose (same dose as before) given 16 weeks later, for a total PfSPZ dose = 22.5 x 10^5. PfSPZ Vaccine administered by DVI.
  Protective efficacy assessed by heterologous CHMI (7G8) Pf parasites at 28 and 40 weeks after the first immunization, along with 8 infectivity controls. Subjects may proceed to CHMI if they have received at least 2 of 4 priming immunizations and the boost scheduled for Group 1. Participants not protected after the first CHMI will be invited to receive a booster vaccination (4.5 x 10^5 PfSPZ) 21 days prior to the second CHMI. Subjects may participate in the second CHMI whether or not they were protected in the 1st CHMI, to serve as controls for the effect of the 1st CHMI on immunity.
  Subjects will be followed for 56 days beyond the final CHMI (post-immunization week 40).
  Interventions: Biological: PfSPZ Vaccine; Biological: CHMI (7G8)
- Group 2 (Experimental): Subjects (n=15) will receive 3 doses of PfSPZ Vaccine (9.0 x 10^5 PfSPZ/dose) every 8 weeks, total PfSPZ dose = 27 x 10^5. PfSPZ Vaccine administered by DVI.
  Protective efficacy assessed by heterologous CHMI (7G8) Pf parasites at 28 and 40 weeks after first immunization, along with 8 infectivity controls. Subjects may proceed to CHMI if they have received at least 2 of 3 immunizations scheduled for Group 2. Participants not protected after the first CHMI will be invited to receive a booster vaccination (9.0 x 10^5 PfSPZ) 21 days prior to the second CHMI. Subjects may participate in the second CHMI whether or not they were protected in the 1st CHMI, to serve as controls for the effect of the 1st CHMI on immunity.
  Subjects will be followed for 56 days beyond the final CHMI (post-immunization week 40).
  Interventions: Biological: PfSPZ Vaccine; Biological: CHMI (7G8)
- Group 3 (Experimental): Group 3 subjects (n=15) will receive 3 doses of PfSPZ Vaccine (18 x 10^5 PfSPZ/dose) every 8 weeks for a total PfSPZ dose of 54 x 10^5. PfSPZ Vaccine administered by DVI.
  Protective efficacy assessed by CHMI with heterologous (7G8, NF135.C10) Pf parasites at 40 and 66 weeks after the first immunization, along with 8 infectivity controls. Subjects may proceed to CHMI if they have received at least 2 of 3 immunizations scheduled for Group 3. All participants will be invited to receive a booster vaccination (18 x 10^5 PfSPZ) 21 days prior to the second CHMI. Subjects may participate in the second CHMI whether or not they were protected in the 1st CHMI, to serve as controls for the effect of the 1st CHMI on immunity.
  Subjects will be followed for 56 days beyond the final CHMI (post-immunization week66).
  Interventions: Biological: PfSPZ Vaccine; Biological: CHMI (7G8); Biological: CHMI (NF135.C10)
- Group 4 (Experimental): Subjects (n=15) will receive a single, priming dose of PfSPZ Vaccine (27 x 10^5 PfSPZ/dose), followed by 2 additional immunizations (9.0 x 10^5 PfSPZ per dose) every 8 weeks, total PfSPZ dose = 45 x 10^5. PfSPZ Vaccine administered by DVI.
  Protective efficacy assessed by CHMI with heterologous 7G8 and NF135.C10 Pf parasites at 40 and 66 weeks, respectively, along with 8 infectivity controls at each CHMI. Subjects may proceed to CHMI if they have received at least 2 of 3 immunizations scheduled for Group 4. All participants will be invited to receive a booster vaccination (9.0x10^5 PfSPZ) 21 days prior to the second CHMI.
  Subjects will be followed for 56 days beyond the final CHMI at (post-immunization week 66).
  Interventions: Biological: PfSPZ Vaccine; Biological: CHMI (7G8); Biological: CHMI (NF135.C10)
- Infectivity Controls, CHMI (7G8) (Other): Infectivity controls (n=24) will not receive any PfSPZ Vaccine. They will serve as infectivity controls for CHMI for all groups. 8 infectivity controls will undergo CHMI with each of two CHMIs (at 28 and 40) for Groups 1 and 2, and 8 infectivity controls will undergo CHMI with the 40 week CHMI for Groups 3 and 4. All CHMI will be conducted by exposure to the bites of 5 mosquitoes infected with heterologous (7G8) Pf parasites. Subjects will be followed for 56 days beyond the last CHMI at week 40 at the UMB site.
  Interventions: Biological: CHMI (7G8)
- Infectivity Controls, CHMI (NF135.C10) (Other): Infectivity controls (n=8) will not receive any PfSPZ Vaccine. They will serve as infectivity controls for the second CHMI at week 66 for Groups 3 and 4. CHMI will be conducted by exposure to the bites of 3-5 mosquitoes infected with heterologous (NF135.C10) Pf parasites. Subjects will be followed for 56 days beyond the last CHMI at week 66 at the NMRC site.
  Interventions: Biological: CHMI (NF135.C10)

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, cryopreserved, radiation-attenuated, Plasmodium falciparum (Pf) sporozoites
  Arms: Group 1; Group 2; Group 3; Group 4
Biological: CHMI (7G8) — CHMI is conducted by exposure to the bites of five mosquitoes infected with heterologous (7G8) Pf parasites.
  Arms: Group 1; Group 2; Group 3; Group 4; Infectivity Controls, CHMI (7G8)
Biological: CHMI (NF135.C10) — CHMI is conducted by exposure to the bites of three to five mosquitoes infected with heterologous (NF135.C10) Pf parasites.
  Arms: Group 3; Group 4; Infectivity Controls, CHMI (NF135.C10)

SUMMARY:
This is an open-label evaluation of the safety, tolerability, immunogenicity and efficacy of PfSPZ Vaccine administered by direct venous inoculation (DVI) in healthy, malaria-naïve adult subjects.

DETAILED DESCRIPTION:
The study will be conducted as a collaborative effort between the NMRC, UMB CVD, WRAIR and Sanaria, Inc. The study screening, immunizations, and follow-ups for Groups 1 & 2 will take place at the UMB CVD. The study screening, immunizations, and follow-ups for Groups 3 & 4 will take place at the NMRC CTC in Bethesda, MD. The controlled human malaria infections (CHMI) will be conducted at WRAIR Entomology, Silver Spring, MD for NMRC subjects, and at UMB CVD for UMB CVD subjects.

There will be 4 groups and a total of 92 subjects (60 immunized subjects and 32 infectivity controls). Group 1 (n = 15) subjects will receive PfSPZ Vaccine administered by direct venous inoculation (DVI), with 4 doses of 4.5 x 10^5 PfSPZ given every two days, followed by a single, boosting dose of 4.5 x 10^5 PfSPZ given 16 weeks later. For participants who were not protected after the first CHMI, an additional boosting dose of 4.5x10^5 PfSPZ will be given 21 weeks later.

Group 2 (n = 15) subjects will receive PfSPZ Vaccine administered by DVI, with 3 doses of 9.0 x 10^5 PfSPZ administered every 8 weeks. For participants who were not protected after the first CHMI, a boosting dose of 9.0 x 10^5 PfSPZ will be given 21 weeks later.

Group 3 (n = 15) subjects will receive PfSPZ Vaccine administered by DVI, with 3 doses of 18 x 10^5 PfSPZ administered every 8 weeks. Following CHMI at 40 weeks, protected subjects and one-half of unprotected subjects will receive a final, boosting dose of 18 x 10^5 PfSPZ. The remaining half of unprotected subjects will receive a final, boosting dose of 4.5 x 10^5 PfSPZ.

Group 4 (n = 15) subjects will receive PfSPZ Vaccine administered by DVI, with 27 x 10^5 PfSPZ administered once as a priming dose, followed by 2 doses of 9.0 x 10^5 PfSPZ administered every 8 weeks. Following CHMI at 40 weeks, protected subjects and one-half of unprotected subjects will receive a final, boosting dose of 9 x 10^5 PfSPZ. The remaining half of unprotected subjects will receive a final, boosting dose of 2.25 x 10^5 PfSPZ.

Protective efficacy will be assessed by CHMI, conducted by exposure to the bites of three to five mosquitoes infected with heterologous (7G8 or NF135.C10) Pf parasites, with the number of mosquitoes depending on the infection intensity in the mosquitoes). At UMB CVD, protective efficacy will be assessed at both 28 and 40 weeks after the first immunization, in Groups 1 and 2, along with 8 infectivity controls for each CHMI. At NMRC, protective efficacy will be assessed at 40 weeks (7G8 infected mosquitoes), and 66 weeks (NF135.C10 infected mosquitoes) after the first immunization, in Groups 3 and 4. Unprotected subjects in Groups 1 and 2, and all subjects in Groups 3 and 4, will be invited to receive a booster vaccination 21 days prior to the second CHMI at the respective sites, in order to assess the efficacy of a booster dose in previously vaccinated persons. These vaccine subjects may participate in the second CHMI whether or not they were protected in the first CHMI, and independent of their decision to receive the booster immunization, to serve as controls for the effect of the first CHMI on immunity. Subjects may proceed to CHMI provided they have received at least two of the three immunizations scheduled for Groups 2-4, or at least two of the four priming immunizations as well as the boost scheduled for Group 1. 7G8-infected mosquitoes may be substituted for NF135.C10 mosquitoes in case of difficulties with mosquito production.

Two subjects in each group will serve as "pilot subjects" in the event of first in human dosing, and will be immunized approximately 24 hours prior to the rest of the subjects in the respective group. If there are no safety concerns identified in the pilot subjects that trigger the stopping rules, then the remainder of subjects will be immunized the day after the pilot subjects are immunized. Subjects will be followed for 56 days beyond both the week 40 and week 66 CHMIs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant female) 18 - 50 years of age, inclusive.
* Able and willing to participate for the duration of the study.
* Able and willing to provide written (not proxy) informed consent.
* Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) ≤35 for vaccine groups or BMI ≤40 for control groups.
* Women of childbearing potential must agree to use effective means of birth control (e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) during the entire study. Women with a history of surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other) must provide written documentation of infertility from a health care provider.
* Willing to refrain from blood donation for 3 years following CHMI.
* Agree not to travel to a malaria endemic region during the entire course of the trial.

Exclusion Criteria:

* Any history of malaria infection, or travel to a malaria endemic region within 6 months prior to first immunization.
* History of long-term residence (>5 years) in area known to have significant transmission of P. falciparum.
* Body weight equal to, or less than, 110 pounds.
* Has evidence of increased cardiovascular disease risk (defined as > 10%, 5 year risk) as determined by the method of Gaziano [Gaziano, 2008]. Risk factors include sex, age, systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/mm2), and reported diabetes status.
* Positive HIV, HBsAg or HCV serology.
* Positive sickle cell screening test.
* An abnormal electrocardiogram, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* Current use of systemic immunosuppressant pharmacotherapy.
* Current significant medical condition (cardiovascular, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination.
* History of a splenectomy.
* History of neurologic disorder (including seizures) or diagnosis of migraine headache.
* History of psychiatric disorders (such as personality disorders, anxiety disorders, or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult.
* Plan for surgery between enrollment and CHMI.
* Females who are pregnant or nursing, females who plan on becoming pregnant or plan to nurse during the study period.
* Known allergy to any component of the vaccine formulation, history of anaphylactic response to mosquito-bites, or any history of anaphylactic reaction, retinal or visual field changes, or known allergy to anti-malarials including chloroquine phosphate, atovaquone/proguanil (Malarone®), or artemether/lumefantrine (Coartem®).
* Receipt of another investigational vaccine or drug within 30 days prior to the first immunization, or plan to participate in another investigational vaccine/drug research during or within 1 month following participation in this study (vaccine recipients).
* Receipt of another investigational vaccine or drug within 30 days prior to CHMI, or plan to participate in another investigational vaccine/drug research during or within 1 month following participation in this study (infectivity controls).
* Receipt of more than three other vaccines during the period 60 days prior to the screening visit to 1 month following participation in this study.
* Personal beliefs that prohibit the receiving of vaccine product containing human serum albumin within the diluent (vaccine recipients only).
* Use or planned use of any drug with anti-malarial activity that would coincide with the periods of immunization or CHMI.
* Anticipated use of medications known to cause drug reactions with atovaquone-proguanil (Malarone®), or artemether/lumefantrine (Coartem®) such as cimetidine, metoclopramide, antacids, and kaolin.
* History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events | 52 weeks
  Incidence and type of adverse events (including breakthrough infections), vital signs, clinical laboratory assessments, physical examination findings post first immunization onwards.
Efficacy | 28 days post-CHMI
  Evidence of vaccine-mediated protection against CHMI at 28 and 40 weeks in Groups 1 and 2 by preventing blood stage infection for 28 days (as detected by qPCR) following CHMI.
  Evidence of vaccine-mediated protection against CHMI at 40 and 66 weeks in Groups 3 and 4 by preventing blood stage infection for 28 days (as detected by blood smear analysis) following CHMI.
Immunological response | 2 weeks post-immunization and 28 days post-CHMI
  Antibody responses by PfCSP ELISA two weeks after the second, third and booster immunizations (Groups 2-4) or after the fourth, fifth and booster immunizations (Group 1) (serum dilution at which the optical density is 1.0 referred to as the OD 1.0)
  Positive predictive values for anti-PfCSP antibody responses at or above a threshold for predicting sterile protection following CHMI (threshold = OD 1.0 of 2,000)

SECONDARY OUTCOMES:
Immunological outcomes | Day of immunization till 28 days post-CHMI
  1. Antibody titers to other Pf proteins by ELISA
  2. Antibody titers to Pf parasite stages by IFA
  3. Capacity of sera from immunized volunteers to inhibit sporozoite invasion (ISI) of hepatocytes in vitro by ISI assay
  4. Analysis of antibodies to any of the thousands of proteins in the Pf proteome using proteome array chips
  5. Analysis of cellular immune responses against PfSPZ, Pf-infected erythrocytes and/or synthetic peptides and/or recombinant proteins from defined Pf proteins by multi-parameter intracellular staining (ICS) by flow cytometry
  6. Analysis of cellular immune responses against PfSPZ, Pf-infected erythrocytes and/or synthetic peptides and/or recombinant proteins from defined Pf proteins by fluorospot assays
  7. Human gene expression profiling focusing on immune response genes
  8. Analysis of host cellular, cytokine and other host responses by Luminex or Luminex-type assays

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Singer, MD, Principal Investigator — Naval Medical Research Center
Locations (2):
- United States (2):
  - University of Maryland-Baltimore, Center for Vaccine Development, Baltimore, Maryland
  - Naval Medical Research Center, Silver Spring, Maryland

REFERENCES:
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Epstein JE, Tewari K, Lyke KE, Sim BK, Billingsley PF, Laurens MB, Gunasekera A, Chakravarty S, James ER, Sedegah M, Richman A, Velmurugan S, Reyes S, Li M, Tucker K, Ahumada A, Ruben AJ, Li T, Stafford R, Eappen AG, Tamminga C, Bennett JW, Ockenhouse CF, Murphy JR, Komisar J, Thomas N, Loyevsky M, Birkett A, Plowe CV, Loucq C, Edelman R, Richie TL, Seder RA, Hoffman SL. Live attenuated malaria vaccine designed to protect through hepatic CD8(+) T cell immunity. Science. 2011 Oct 28;334(6055):475-80. doi: 10.1126/science.1211548. Epub 2011 Sep 8. PMID 21903775
- [Background] Ishizuka AS, Lyke KE, DeZure A, Berry AA, Richie TL, Mendoza FH, Enama ME, Gordon IJ, Chang LJ, Sarwar UN, Zephir KL, Holman LA, James ER, Billingsley PF, Gunasekera A, Chakravarty S, Manoj A, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, K C N, Murshedkar T, DeCederfelt H, Plummer SH, Hendel CS, Novik L, Costner PJ, Saunders JG, Laurens MB, Plowe CV, Flynn B, Whalen WR, Todd JP, Noor J, Rao S, Sierra-Davidson K, Lynn GM, Epstein JE, Kemp MA, Fahle GA, Mikolajczak SA, Fishbaugher M, Sack BK, Kappe SH, Davidson SA, Garver LS, Bjorkstrom NK, Nason MC, Graham BS, Roederer M, Sim BK, Hoffman SL, Ledgerwood JE, Seder RA. Protection against malaria at 1 year and immune correlates following PfSPZ vaccination. Nat Med. 2016 Jun;22(6):614-23. doi: 10.1038/nm.4110. Epub 2016 May 9. PMID 27158907
- [Background] Lyke KE, Ishizuka AS, Berry AA, Chakravarty S, DeZure A, Enama ME, James ER, Billingsley PF, Gunasekera A, Manoj A, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Kc N, Murshedkar T, Mendoza FH, Gordon IJ, Zephir KL, Holman LA, Plummer SH, Hendel CS, Novik L, Costner PJ, Saunders JG, Berkowitz NM, Flynn BJ, Nason MC, Garver LS, Laurens MB, Plowe CV, Richie TL, Graham BS, Roederer M, Sim BK, Ledgerwood JE, Hoffman SL, Seder RA. Attenuated PfSPZ Vaccine induces strain-transcending T cells and durable protection against heterologous controlled human malaria infection. Proc Natl Acad Sci U S A. 2017 Mar 7;114(10):2711-2716. doi: 10.1073/pnas.1615324114. Epub 2017 Feb 21. PMID 28223498
- [Background] Epstein JE, Paolino KM, Richie TL, Sedegah M, Singer A, Ruben AJ, Chakravarty S, Stafford A, Ruck RC, Eappen AG, Li T, Billingsley PF, Manoj A, Silva JC, Moser K, Nielsen R, Tosh D, Cicatelli S, Ganeshan H, Case J, Padilla D, Davidson S, Garver L, Saverino E, Murshedkar T, Gunasekera A, Twomey PS, Reyes S, Moon JE, James ER, Kc N, Li M, Abot E, Belmonte A, Hauns K, Belmonte M, Huang J, Vasquez C, Remich S, Carrington M, Abebe Y, Tillman A, Hickey B, Regules J, Villasante E, Sim BKL, Hoffman SL. Protection against Plasmodium falciparum malaria by PfSPZ Vaccine. JCI Insight. 2017 Jan 12;2(1):e89154. doi: 10.1172/jci.insight.89154. PMID 28097230
- [Derived] Lyke KE, Singer A, Berry AA, Reyes S, Chakravarty S, James ER, Billingsley PF, Gunasekera A, Manoj A, Murshedkar T, Laurens MB, Church WP, Garver Baldwin LS, Sedegah M, Banania G, Ganeshan H, Guzman I, Reyes A, Wong M, Belmonte A, Ozemoya A, Belmonte M, Huang J, Villasante E, Sim BKL, Hoffman SL, Richie TL, Epstein JE; Warfighter II Study Team. Multidose Priming and Delayed Boosting Improve Plasmodium falciparum Sporozoite Vaccine Efficacy Against Heterologous P. falciparum Controlled Human Malaria Infection. Clin Infect Dis. 2021 Oct 5;73(7):e2424-e2435. doi: 10.1093/cid/ciaa1294. PMID 32920641